CLINICAL TRIAL: NCT00557492
Title: Phase II Study of the Anti-Vascular Endothelial Growth Factor (α-VEGF) Monoclonal Antibody Bevacizumab in Combination With Fixed Dose Rate (FDR) Gemcitabine and Rapid-Fractionation Radiotherapy in the Pre-operative Treatment of Potentially- Resectable Pancreatic Adenocarcinoma
Brief Title: Efficacy of Neoadjuvant Chemoradiation for Potentially Resectable Pancreas Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amer Zureikat (Other)
Responsible Party: Sponsor-Investigator, Amer Zureikat, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-035; NCT00428324 (obsolete NCT alias)
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Pancreatic Cancer
Keywords: pancreas; pancreatic; cancer; resectable
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Bevacizumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Intervention: Drug: Avastin (bevacizumab) 10 mg/kg, days 1, 15, 29 and 43
  Intervention: Drug: Gemzar (Gemcitabine) On days 1, 15, and 29, subjects will receive gemcitabine 1500 mg/m2 IV over 150 minutes at the fixed-dose rate (10 mg/m2/min).
  Intervention:Radiation: external beam radiotherapy 3 Gy/fraction utilizing a 95% isodose field over 10 consecutive weekdays, Monday to Friday, for a total of 30 Gy
  Interventions: Drug: Avastin (bevacizumab); Drug: Gemzar (Gemcitabine); Radiation: external beam radiotherapy

INTERVENTIONS:
Drug: Avastin (bevacizumab) — 10 mg/kg, days 1, 15, 29 and 43
Drug: Gemzar (Gemcitabine) — On days 1, 15, and 29, subjects will receive gemcitabine 1500 mg/m2 IV over 150 minutes at the fixed-dose rate (10 mg/m2/min).
Radiation: external beam radiotherapy — 3 Gy/fraction utilizing a 95% isodose field over 10 consecutive weekdays, Monday to Friday, for a total of 30 Gy

SUMMARY:
This study is to determine the efficacy of bevacizumab and gemcitabine in combination with radiation therapy in the preoperative treatment of potentially-resectable subjects with pancreatic cancer.

DETAILED DESCRIPTION:
This is a 2 stage phase II study of bevacizumab (10 mg/kg) and fixed dose rate (FDR) gemcitabine (1500 mg/m2 at 10 mg/kg/min) in combination with sequential rapid fractionation radiotherapy (30 Gy total) in the preoperative treatment of potentially-resectable subjects with adenocarcinoma of the pancreas. The purpose of this study is to determine the rate of margin negative surgical resection (R0 resection rate) and the rate of complete pathological response in patients with resected pancreas cancer. The overall goal of this study is to determine the merit of this novel regimen for further study in a Phase III trial examining time to progression and overall survival. Based on the need for 48 evaluable subjects to evaluate the primary endpoints, the study will be opened with a target accrual of 60 subjects given an expected 20% rate of attrition observed in prior studies of subjects with pancreas cancer at UPCI.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic proof of pancreatic adenocarcinoma.
* Subjects with biopsy-proven adenocarcinoma of the pancreas which is potentially resectable by preoperative imaging. Subjects will be considered potentially resectable using criteria defined by Pisters (Pisters et al., 2001):
* if imaging detects no evidence of extrapancreatic disease;
* no evidence of tumor extension to the superior mesenteric artery (SMA) or celiac axis (intact fat plane between the tumor and the adjacent visceral artery),
* patent superior mesenteric-portal vein confluence
* no encasement of portal or superior mesenteric vein.
* Karnofsky performance status ≥ 80.
* No active second malignancy except for basal cell carcinoma of the skin
* Normal renal, hepatic, and hematologic function at the time of enrollment as evidenced by:
* Serum creatinine level ≤1.6 mg/dl ( Calculated Creat clearance >50)
* Serum total bilirubin level ≤1.5 X ULN
* Urine protein excretion ≤ 1+ by urine dipstick
* White blood cell count ≥ 3.5x109/ml per ml and platelet count ≥ 100x109 per ml
* Age >18 years.
* Children are excluded because of toxic effects of bevacizumab and gemcitabine on growth and development during preclinical studies.
* For subjects with obstructive jaundice, the biliary tract must be drained with a temporary plastic or a short permanent metallic biliary stent.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Disease-Specific Exclusions
* Subjects who have received chemotherapy within 12 months prior to study entry.
* Prior use of radiotherapy or investigational agents for pancreatic cancer.
* Subjects who have undergone laparotomy for pancreas cancer within 6 weeks
* Any evidence of metastasis to distant organs (liver, lung, peritoneum).
* Symptomatic or endoscopic evidence of gastric outlet obstruction

  • Endoscopic findings suggesting tumor erosion into the gastrointestinal mucosa.
* Concurrent malignancies with evidence of active or measurable disease except basal cell carcinoma of the skin.
* General Medical Exclusions
* Inability to adhere to study and/or follow-up procedures
* History of allergic reactions or hypersensitivity to the study drugs (bevacizumab, gemcitabine, and proton pump inhibitors).
* Other concurrent experimental therapy.
* Because subjects with immune deficiency are at increased risk for lethal infections when treated with marrow-suppressive therapy, HIV-positive subjects receiving combination anti-retroviral therapy are excluded from the study.
* Bevacizumab-Specific Exclusions
* Subjects who have had recent surgery (prior 6 weeks)
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* Subjects with the following co-morbid medical conditions:
* History of myocardial infarction or unstable angina within 12 months prior to study enrollment.
* Ascites
* Pregnancy/lactation - The effects of the study drugs on the developing human fetus are unknown. For this reason and because bevacizumab, gemcitabine, and radiation therapy used in this trial are known to be teratogenic in animal studies, women and men of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from the time of study entry until 6 months after the completion of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A serum pregnancy test for those females of childbearing potential must be done prior to their receiving study drugs. Due to the combined effects of chemotherapy and radiation, breastfeeding is not allowed for 6 months after the completion of study participation.
* Regular aspirin use > 325 mg per day
* Regular NSAID use
* Bleeding diathesis, coagulopathy, need for full-dose anticoagulation or INR > 1.5
* Known central nervous system metastasis
* Previous cerebrovascular accident, transient ischemic attack, or seizure (within 6 months)
* Serious non-healing wound, ulcer, or bone fracture
* History of abdominal fistula, gastrointestinal perforation, diverticulitis, or intra-abdominal abscess within 6 months prior to study enrollment.
* Recent hemoptysis,
* Uncontrolled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) grade 2 or greater congestive heart failure (see Appendix I)
* Prior deep venous thrombosis or pulmonary embolism
* Urine protein excretion 2+ or ≥ 1 g per 24 hours
* Peripheral vascular disease such as lower extremity claudication and rest pain or prior lower extremity vascular surgery for arterial insufficiency
* Dyspnea requiring supplemental oxygen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-12; Primary Completion 2012-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert J. Zeh, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Centers, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FDR GEM + BEV +/- BEV/RT: Participants received fixed-dose rate (FDR) gemcitabine (GEM) (1,500 mg/m^2) plus bevacizumab (BEV) (10 mg/kg IV) every 2 weeks for three cycles followed by accelerated RT (30 Gy in 10 fractions) plus BEV directed at gross tumor volume plus a 1-2 cm vascular margin, +/- laparoscopy and resection after day 85.
Period: Overall Study
Arm/Group | FDR GEM + BEV +/- BEV/RT
Started | 59
Completed | 58 (Evaluable for outcomes)
Not Completed | 1
Not completed — Change in health insurance | 1

BASELINE CHARACTERISTICS:
Arm/Group | FDR GEM + BEV +/- BEV/RT
Number analyzed (Participants) | 59
Age, Continuous [Median (Full Range); unit: years] | 60 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Rate of Margin Negative Surgical Resection (R0 Resection Rate)
Description: Number of participants who underwent laparoscopy and pancreatic resections that were margin negative/total number of participants who underwent laparoscopy and pancreatic resections.
Time Frame: Up to 48 months
Population: Participants who underwent laparoscopy and pancreatic resection.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FDR GEM + BEV +/- BEV/RT
Number analyzed (Participants) | 43
percentage of participants | 88 [75 to 96]

2. Primary Outcome: Rate of Pathologic Complete Response (pCR)
Description: Rate of pathologic complete response (pCR) is no residual invasive tumor, in situ carcinoma can be present, and no residual lymph node metastasis. Rate of pCR is the number of participants who underwent laparoscopy and pancreatic resections that experienced complete pathologic response/total number of participants who underwent laparoscopy and pancreatic resections.
Time Frame: Up to 48 months
Population: Participants who underwent laparoscopy and pancreatic resections.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FDR GEM + BEV +/- BEV/RT
Number analyzed (Participants) | 43
percentage of participants | 2.3 [0.1 to 12]

3. Secondary Outcome: Overall Survival (OS)
Time Frame: Up to 48 months
Population: Includes entire study cohort.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | FDR GEM + BEV +/- BEV/RT
Number analyzed (Participants) | 58
months | 16.8 [14.9 to 21.3]

4. Secondary Outcome: Overall Survival (OS)
Time Frame: Up to 48 months
Population: Includes participants who underwent laparoscopy and pancreatic resection.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | FDR GEM + BEV +/- BEV/RT
Number analyzed (Participants) | 43
months | 19.7 [16.5 to 28.2]

5. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: Up to 48 months
Population: Includes entire study cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FDR GEM + BEV +/- BEV/RT
Number analyzed (Participants) | 58
months | 6.6 [4.9 to 12.4]

6. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: Up to 48 months
Population: Includes participants who underwent laparoscopy and pancreatic resection.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FDR GEM + BEV +/- BEV/RT
Number analyzed (Participants) | 43
months | 12.9 [7.0 to 18.7]

7. Secondary Outcome: Rate of Surgical Resection
Description: Number of participants that underwent resection / per the total number of evaluable participants
Time Frame: Up to 48 months
Measure: Number; unit: percentage of participants
Arm/Group | FDR GEM + BEV +/- BEV/RT
Number analyzed (Participants) | 58
percentage of participants | 74

8. Secondary Outcome: Radiographic Tumor Response
Description: CT scans evaluated for response using Response Evaluation Criteria in Solid Tumors (RECIST)
Time Frame: Up to 48 months
Measure: Number; unit: Participants
Arm/Group | FDR GEM + BEV +/- BEV/RT
Number analyzed (Participants) | 58
Participants
  metastatic progression (at restaging) | 4
  stable disease | 39
  partial response | 5
  progressive disease | 10

9. Secondary Outcome: Ca 19-9 Level (in Serum) - Biomarker Response
Description: Percentage decrease in Ca 19-9 level (in serum)
Time Frame: Baseline and up to 48 months
Population: Participants that did NOT demonstrate metastatic progression upon restaging CT.
Measure: Mean (Standard Deviation); unit: percentage decrease in serum Ca19-9 leve
Arm/Group | FDR GEM + BEV +/- BEV/RT
Number analyzed (Participants) | 54
percentage decrease in serum Ca19-9 leve | 25 (80)

ADVERSE EVENTS:
Arm/Group | FDR GEM + BEV +/- BEV/RT
Serious Adverse Events (participants affected / at risk) | 10/59
Other Adverse Events (participants affected / at risk) | 50/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FDR GEM + BEV +/- BEV/RT (N=59)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Leak (including anastomotic), GI, Pancreas (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Obstruction, GI, Small bowel NOS (Gastrointestinal disorders) | 1
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 1
Hepatobiliary/Pancreas (Hepatobiliary disorders) | 1
Infection (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Abdomen NOS (Infections and infestations) | 2
Pain, Abdomen NOS (General disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FDR GEM + BEV +/- BEV/RT (N=59)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 5
Platelets (Blood and lymphatic system disorders) | 7
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 8
Hemoglobin (Blood and lymphatic system disorders) | 9
Fatigue (asthenia, lethargy, malaise) (General disorders) | 21
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 4
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 6
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 6
Gastrointestinal (Gastrointestinal disorders) | 6
Anorexia (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 21
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 7
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 8
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 9
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 9
Alkaline phosphatase (Metabolism and nutrition disorders) | 11
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 13
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 16
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 22
Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 4
Mood alteration, Anxiety (Nervous system disorders) | 6
Pain (General disorders) | 5
Pain, Head/headache (General disorders) | 6
Pain, Abdomen NOS (General disorders) | 12
Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes